CLINICAL TRIAL: NCT06337799
Title: Use of Non-physician Allied-health Professionals to Recruit (and Follow) Research Participants, Sustain Engagement, and Improve and Diagnose Treatment of Diseases by Facilitating Transitions of Care
Brief Title: Use of Allied-health Professionals to Improve Treatment of Disease
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Philip Polgreen, Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202210411
Record Dates: First submitted 2024-03-22; First posted 2024-03-29 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Preeclampsia
MeSH Terms: conditions — Pre-Eclampsia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Research Pharmacist Monitoring (Experimental): The research pharmacist will help the mother find a primary care physician if she doesn't have one and discuss strategies to lower blood pressure, if needed. The pharmacist interactions will occur 7 days after enrollment and then approximately every 2 weeks to 2 months during 12 months of follow up, depending on blood pressure control. They may recommend medications to the participant's physician. The pharmacist will have access to the participant's electronic medical record to obtain any blood pressure-related medications that the mother is prescribed as well as throughout the follow up to ensure any health-related conditions can be discussed.
  Interventions: Behavioral: Research Pharmacist

INTERVENTIONS:
Behavioral: Research Pharmacist — The goal of this intervention is to determine if allied health professionals will improve blood pressure in new mothers.

SUMMARY:
The goal of this clinical trial is to learn if allied-health professionals can recruit and follow research participants, sustain engagement, and improve and diagnose treatment of diseases by facilitating transitions of care.

Participants will:

Take their blood pressure at home and return it to the research team; Follow up with a research pharmacist for 12 months; Return for a follow up visit after 12 months.

DETAILED DESCRIPTION:
After consent, a research pharmacist will virtually monitor the participant's blood pressure until the 12-month follow up visit. The research pharmacists will have access to the participant's electronic medical records to monitor and document medications and clinic blood pressures for analysis . Participants will be asked to measure and return 14 blood pressure measurements (2x per day for 7 days) using our text messaging platform. They will be allowed to choose the times that they are sent reminders to measure their blood pressure. If a participant has blood pressure values sufficient for a hypertension diagnosis, the pharmacist will communicate via electronic medical record with the participant's primary care team. If they do not have a primary care provider, the pharmacist will facilitate finding one. The pharmacist will continue monitoring the participant and making recommendations to the primary care team through the electronic medical record to quickly adjust therapy to improve blood pressure control. The pharmacists will typically contact the participants (via participant's choice of phone, text, or email) every 2-3 weeks while their hypertension is uncontrolled. Once under control, the pharmacist will continue to contact the participant at least every 2 months to support adherence and reassess control.

ELIGIBILITY:
Inclusion Criteria:

* Biological mothers delivering at UIHC or attending a well-child visit for an infant between 1 month and 9 months
* Preeclampsia during pregnancy
* Preceived prenatal care at UIHC
* Owns a smartphone

Exclusion Criteria:

* Arm circumference greater than 17 inches
* Prisoner status
* Unable to provide own written informed consent

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 200 (Estimated)
Dates: Start 2026-10 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Number of Subjects at Risk for Hypertension | Through study completion, an average of 12 months
  We will calculate the number of participants who are at risk for hypertension during the course of the intervention.
Number of Subjects Exposed to a Screening Clinic | Through study completion, an average of 12 months
  We will calculate the number of participants who visited a screening clinic during the course of the intervention.
Number of Subjects Screened at a Screening Clinic | Through study completion, an average of 12 months
  We will calculate the number of participants who were screened at a screening clinic during the intervention.
Number of Subjects Followed-Up by the Research Pharmacist | Through study completion, an average of 12 months
  We will calculated the number of participants who were followed-up by a research pharmacist during the intervention.
Number of Subjects Diagnosed with Hypertension | Through study completion, an average of 12 months
  We will calculate the number of participants who were diagnosed with hypertension by their provider during the intervention.
Number of Subjects Treated for Hypertension, if Diagnosed | Through study completion, an average of 12 months
  We will calculate the number of participants who were treated for their hypertension diagnosis by their provider, if they were diagnosed with hypertension, during the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Philip M Polgreen, MD, Principal Investigator — University of Iowa